CLINICAL TRIAL: NCT06954493
Title: Phase 1, Open-Label Pharmacokinetic Study in Healthy Lactating Women After Two Oral Doses of Ibrexafungerp Administered on a Single Day
Brief Title: Pharmacokinetic Study in Healthy Lactating Women Exposed to Ibrexafungerp
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scynexis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCY-078-121
Record Dates: First submitted 2024-01-09; First posted 2025-05-01 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-04

CONDITIONS: Vulvovaginal Candidiasis; Candida Infection; Vaginal Candidiasis
Keywords: VVC; Thrush; BREXAFEMME; Candidiasis; Vaginal Yeast; Yeast Infection; Lactating; Fungal Disease; Fungal Infection
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Candidiasis; Candidiasis, Oral; Mycoses | interventions — ibrexafungerp

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label Treatment (Other): Participants received a single day of twice daily (BID) 300-mg (2 x 150-mg) oral ibrexafungerp doses given 12 hours apart (Q12H)
  Interventions: Drug: Ibrexafungerp

INTERVENTIONS:
Drug: Ibrexafungerp — Ibrexafungerp Oral Tablet

SUMMARY:
This is a pharmacokinetic evaluation of lactating women after receiving two doses of Ibrexafungerp. The study population included healthy lactating females who were at least 10 days postpartum with a fully established milk supply and were between the ages of 18 and 50 years at the time of screening

DETAILED DESCRIPTION:
This was a Phase 1 study designed to evaluate the pharmacokinetics of ibrexafungerp after administration of two oral doses in lactating women to determine whether ibrexafungerp is excreted in breast milk, and if so, to characterize ibrexafungerp PK in the breast milk and plasma of lactating women.

Participants received a single day of twice daily (BID) 300-mg (2 x 150-mg) oral ibrexafungerp doses given 12 hours apart (Q12H). Participants received both doses on site. Participants were admitted to the clinic on Day 1 and discharged on Day 5, after the 108-hour procedures were completed.

ELIGIBILITY:
Inclusion Criteria:

* A healthy lactating woman aged 18 to 50 years, inclusive, at Screening
* At least 10-days postpartum after uncomplicated delivery with a full milk supply established. (There is no specific length of time postpartum)
* Actively breastfeeding or expressing breast milk
* willing to temporarily discontinue breast feeding their infant before the Day 1 morning dose through to 108 hours after the first dose (approximately 4.5 days) AND has the ability to pump breast milk and to provide a reserve for infant feeding, with acceptance of bottle feeding, prior to the study OR has decided to discontinue breastfeeding permanently but has not yet started weaning their infant with acceptance of bottle feeding and must have adequate milk supply
* Has a Body Mass Index (BMI) ≤34 kg/m2 at the screening visit. BMI is calculated by taking the participant's weight in kg and dividing by the participant's height in meters, squared.
* willing to fully express breast milk from both breasts during the duration of the milk collection portion of the study
* Is judged to be in good health based on medical history, physical examination, vital sign measurements, and laboratory safety tests (all within laboratory normal ranges or changes outside the normal range judged to be clinically non-significant by the investigator) performed at the screening visit and prior to administration of the initial dose of study drug
* Has no clinically significant abnormality on electrocardiogram (ECG) performed at the screening visit
* Has been a non-smoker (including vaping) or a light smoker (less than 10 cigarettes per day) for at least 6 months
* Understands the study procedures and agrees to participate in the study by giving written informed consent
* Is willing to comply with the study restrictions and participate for the full length of the study for a complete summary of study restrictions
* Is not pregnant and highly unlikely to become pregnant

Exclusion Criteria:

* Is pregnant or unwilling or unable to comply with the lifestyle guidelines presented in the protocol during the study period and through the Post-Study visit
* Has evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric (including post-natal depression), neurologic, allergic disease (including drug allergies, but excluding untreated asymptomatic, seasonal allergies at time of dosing), or a history of neoplastic disease or any active cancer
* Is mentally or legally incapacitated
* Has a history of any illness or clinical findings that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the participant or infant by participation in the study
* Anticipates the use of prescription or non-prescription drugs that are strong CYP3A4 inducers, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days of study drug administration (or 14 days if the drug is a potential enzyme inducer)
* Is unable to refrain from consumption of grapefruit juice, grapefruits, grapefruit products, star fruit, Seville and blood oranges, apple and mulberry juice as well as vegetables from the mustard green family (eg, kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, and mustard), charbroiled meats, and fenugreek beginning approximately 7 days prior to administration of the initial dose of study drug and throughout the participant's stay in the clinic
* Consumes significant amounts of alcohol, defined as greater than 2 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces] or distilled spirits [25 mL/1 ounce]) per day. Participant is unable to refrain from all alcohol consumption within one week prior to study dosing throughout the study until the final study visit
* Consumes excessive amounts of caffeine for one month prior to study drug administration, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola or other caffeinated beverages per day
* Has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) or participated in another investigational study within 30 days or 5½ half-lives of the investigational product prior to the screening. The 30-day window will be derived from the date of the last study procedure (ie, poststudy, AE follow-up, etc.) in the previous study to the screening visit of the current study
* Has a history of significant multiple and/or severe allergies [including latex allergy, but with exception of seasonal rhinitis (hay fever)] or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Has a known hypersensitivity to ibrexafungerp
* Is currently a user including illicit drugs or has a history of drug (including alcohol) abuse within approximately 1 year
* Is unable to abstain from strenuous exercise from the screening visit until administration of the initial dose of study drug, throughout the study until the poststudy visit

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Lactating women
Enrollment: 5 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Woodland Research Northwest (WRN), Rogers, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is an open-label study.
Groups:
- Open Label Treatment: Participants will receive a single day of twice daily (BID) 300-mg (2 x 150-mg) oral ibrexafungerp doses given 12 hours apart (Q12H)
Period: Overall Study
Arm/Group | Open Label Treatment
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Count of Participants; unit: Participants] — BMI in kg/m^2 taking the subjects weight in kg and dividing it by their height in meters squared.
  Participants
    BMI 15 to <20 | 1
    BMI 20 to <25 | 2
    BMI 25 to <30 | 2

OUTCOME MEASURES:

1. Primary Outcome: SCY-078 Breast Milk Concentrations.
Description: To determine the levels of SCY-078 in breast milk in ng/mL, starting pre-dose (Baseline) on Day 1 until 108 hours post first dose. Concentrations of SCY-078 in milk is measured pre-dose, and in milk collected at the following post-dose intervals: 0-2 hours, 2-4 hours, 4-8 hours, 8-12 hours, 12-18 hours, 18-24 hours, 24-36 hours, 36-48 hours, 48-72 hours and 72-108 hours.
Time Frame: Pre-dose up to 108 hours post first dose
Population: Pharmokinetic Population - all subjects that received ibrexafungerp (SCY-078) and that had at least one quantifiable Pk parameter.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 5
ng/mL
  Pre-dose (Baseline) | 0 [0 to 0]
  0-2 hours | 37.64 [9.8 to 49.8]
  2-4 hours | 72.22 [32.1 to 94.1]
  4-8 hours | 43.85 [36.8 to 84.1]
  8-12 hours | 25.62 [20.1 to 73.9]
  12-18 hours | 44.9 [29.8 to 66.6]
  18-24 hours | 51.87 [42.3 to 65.3]
  24-36 hours | 43.48 [22.7 to 60.6]
  36-48 hours | 13.8 [12.6 to 42.0]
  48-72 hours | 8.04 [7.0 to 22.2]
  72-108 hours | 0.00 [0.0 to 11.0]

2. Primary Outcome: SCY-078 Plasma Concentrations.
Description: To measure the levels of SCY-078 in plasma at pre-dose (0 hours), 2, 6, 8 12 hours post dose (prior to the second dose) and 24, 36, 48, 72 and 108 hours post first dose.
Time Frame: Pre-dose up to 72-108 hours post first dose
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 5
ng/mL
  0 hours | 0 [0 to 0]
  2 hours | 321.25 [256.7 to 556.4]
  6 hours | 437.81 [202.5 to 530.7]
  8 hours | 370.76 [216.3 to 432.1]
  12 hours | 315.17 [153.8 to 333.0]
  24 hours | 400.06 [265.3 to 481.4]
  36 hours | 295.15 [137.8 to 317.1]
  48 hours | 145.12 [72.1 to 195.1]
  72 hours | 59.89 [38.7 to 95.2]
  108 hours | 21.56 [11.4 to 36.9]

3. Secondary Outcome: Potential Infant Exposure
Description: The daily infant dosage (total drug present in milk and potentially consumed by the infant per day) is calculated using the following formula:
  Daily Infant Dosage (mg/day) = Σ (total drug concentration in each milk collection multiplied by the expressed milk volume in each milk collection)
Time Frame: Day 1 of dosing (0-24 hours post dose)
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/day
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 5
mg/day | 0.0303 [0.006 to 0.156]

4. Secondary Outcome: Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Any participant who experiences a Treatment Emergent Adverse Event (TEAE).
Time Frame: From the time of consent up to 108 hours post dose
Population: Safety Population - All participants who were enrolled in the study and received at least a partial tablet of ibrexafungerp.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 5
Participants | 1

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Adverse events are reported for all participants in the study.
Time Frame: From the time of consent up to 108 hours post-dose
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 5
Participants
  Gastrointestinal disorders - Soft Stool | 1
  No TEAEs | 4

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of consent through the End of Study Visit (approximately 5 days)
Arm/Group | Open Label Treatment
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Treatment (N=5)
Faeces soft / SOFT STOOL (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT06954493/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/93/NCT06954493/SAP_001.pdf